CLINICAL TRIAL: NCT03925649
Title: Individual Patient Expanded Access IND (Investigational New Drug) of Autologous HB-adMSCs for the Treatment of Spinal Cord Injury
Brief Title: Individual Patient Expanded Access IND of Hope Biosciences Autologous Adipose-derived Mesenchymal Stem Cells for Treatment of SCI
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences LLC (Industry)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Organization: Hope Biosciences Research Foundation (Industry)
Other Study IDs: HBSCI01
Record Dates: First submitted 2019-04-16; First posted 2019-04-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury at C5-C7 Level
Keywords: SCI; stem cells; quadriplegia; spinal cord injury; paralysis; MSCs
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries; Paralysis

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate, Treatment

INTERVENTIONS:
Biological: HB-adMSCs — single infusion of HB-adMSCs

SUMMARY:
This study is expanded access to an Investigational New Drug (IND) for an individual patient with spinal cord injury (SCI) at cervical spine 5-6 (C 5-6) designed to provide access to autologous adipose-derived mesenchymal stem cells (HB-adMSCs)

DETAILED DESCRIPTION:
This is an expanded access single-dose study with the primary goal of treatment submitted at the request of an individual patient with complete C5-6 spinal cord injury (SCI) resulting in quadriplegia who does not qualify for any current clinical trials and for whom there are no other FDA approved fully restorative treatments. The overall objective of this study is to evaluate patient's response, adverse events and serious adverse events (AE/SAEs), and cell expansion characteristics of a single intravenous (IV) infusion of autologous adipose-derived mesenchymal stem cells (HB-adMSCs) in a subject with complete SCI resulting in quadriplegia.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively intact, capable of giving informed consent
* Clinical diagnosis of a non-penetrating traumatic SCI
* Asia Impairment Scale grade of A, B, or C

Exclusion Criteria:

1. Prior history of:

   * Brain injury
   * Recent or ongoing infection
   * Clinically significant cardiovascular, lung, renal, hepatic or endocrine disease,
   * Neurodegenerative disorders
   * Cancer
   * Immunosuppression as defined by WBC<3,000 cells/ml at baseline screening,
   * HIV+
   * Chemical or ETOH dependency
2. Having a contraindication to MRI scans
3. Other acute or chronic medical conditions that, in the opinion of the investigator, may increase the risks associated with study participation or HB-adMSC administration
4. Participation in other interventional research studies
5. Unwillingness to return for follow-up visits

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Hermann Hospital-Clinical Research Unit (MMH-CRU), Houston, Texas, United States